CLINICAL TRIAL: NCT02012699
Title: Integrated Cancer Repository for Cancer Research
Acronym: iCaRe2
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0253-13-EP; NCT00693368 (obsolete NCT alias)
Record Dates: First submitted 2013-12-02; First posted 2013-12-16 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer; Thyroid Cancer; Lung Cancer; Esophageal Cancer; Thymus Cancer; Colon Cancer; Rectal Cancer; Gastrointestinal Stromal Tumors; Anal Cancer; Bile Duct Cancer; Duodenal Cancer; Gallbladder Cancer; Gastric Cancer; Liver Cancer; Small Intestine Cancer; Peritoneal Surface Malignancies; Familial Adenomatous Polyposis; Lynch Syndrome; Bladder Cancer; Kidney Cancer; Penile Cancer; Prostate Cancer; Testicular Cancer; Ureter Cancer; Urethral Cancer; Hypopharyngeal Cancer; Laryngeal Cancer; Lip Cancer; Oral Cavity Cancer; Nasopharyngeal Cancer; Oropharyngeal Cancer; Paranasal Sinus Cancer; Nasal Cavity Cancer; Salivary Gland Cancer; Skin Cancer; Central Nervous System Tumor; Central Nervous System Cancer; Mesothelioma; Breast Cancer; Leukemia; Melanoma; Sarcoma; Unknown Primary Tumor; Multiple Myeloma; Ovarian Cancer; Endometrial Cancer; Vaginal Cancer; Neuroendocrine Tumors; Plasma Cell Dyscrasia; Healthy Control
Keywords: Pancreatic Cancer; Thyroid Cancer; Esophageal cancer; Thymus cancer; Pancreatic tumor; Esophageal tumor; Thymus tumor; Thyroid Tumor; Thyroid Nodule; Lung Tumor; Breast Cancer; Neuroendocrine tumor; Plasma Cell Dyscrasia; Healthy Control
MeSH Terms: conditions — Pancreatic Neoplasms; Thyroid Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Thymus Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Gastrointestinal Stromal Tumors; Anus Neoplasms; Bile Duct Neoplasms; Duodenal Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Liver Neoplasms; Peritoneal Neoplasms; Adenomatous Polyposis Coli; Colorectal Neoplasms, Hereditary Nonpolyposis; Urinary Bladder Neoplasms; Kidney Neoplasms; Penile Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Ureteral Neoplasms; Urethral Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Lip Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Paranasal Sinus Neoplasms; Salivary Gland Neoplasms; Skin Neoplasms; Central Nervous System Neoplasms; Mesothelioma; Breast Neoplasms; Leukemia; Melanoma; Sarcoma; Neoplasms, Unknown Primary; Multiple Myeloma; Ovarian Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Neuroendocrine Tumors; Paraproteinemias; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Biospecimen Retention: Samples With DNA — Blood: Optional Donation. At enrollment and other time points during routine care visits, typically before or after treatment changes. Approximate amounts are 2 tablespoons and total annual amount will not exceed 20 tablespoons.
  Urine: Optional Donation. At enrollment and follow up appointments, if on active study.
  Tissue: Portion of leftover tissue collected and saved from surgery/biopsy, including,but not limited to tumor tissue and/or metastatic cancer tissue and/or paraffin embedded tissue prospectively or retrospectively collected.
  Questionnaire: Baseline and follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The iCaRe2 is a multi-institutional resource created and maintained by the Fred & Pamela Buffett Cancer Center to collect and manage standardized, multi-dimensional, longitudinal data and biospecimens on consented adult cancer patients, high-risk individuals, and normal controls. The distinct characteristic of the iCaRe2 is its geographical coverage, with a significant percentage of small and rural hospitals and cancer centers. The iCaRe2 advances comprehensive studies of risk factors of cancer development and progression and enables the design of novel strategies for prevention, screening, early detection and personalized treatment of cancer. Centers with expertise in cancer epidemiology, genetics, biology, early detection, and patient care can collaborate by using the iCaRe2 as a platform for cohort and population studies.

DETAILED DESCRIPTION:
The integrated Cancer Repository for Cancer Research (iCaRe2 http://icare2.unmc.edu) is a unique sociotechnical resource for the collection and management of cancer and health-related data at the Fred & Pamela Buffett Cancer Center at University of Nebraska Medical Center (UNMC). The iCaRe2 is a multi-center, semantically interoperable and easily customizable cancer data resource, which is aimed at collecting, managing, mining and sharing the comprehensive, multi-dimensional cancer-related data on cancer patients and biospecimens (such as tumor specimens, germ line DNA, serum, urine, and plasma) collected from those individuals.

The iCaRe2 has been developed as an expansion of the biocomputing framework that initially included four multi-center collaborative registries: Pancreatic Cancer Collaborative Registry (PCCR), Breast Cancer Collaborative Registry (BCCR), Thyroid Cancer Collaborative Registry (TCCR), and Great Plains Health Informatics Database (GPHID; to enroll subjects with no history of cancer diagnosis at time of enrollment). The repository now includes: Thoracic Oncology Collaborative Registry (TOCR), GenitoUrinary Cancer Collaborative Registry (GUCARE), Head and Neck Cancer Collaborative Registry (HNCCR), Gastrointestinal & Abdominal Cavity Cancer Collaborative Registry (GACCaRe), Central Nervous System Tumor Collaborative Registry (CTCR), Leukemia and Myeloid Neoplasm Registry (LEMN) , Gynecological Cancer Collaborative Registry (GCCR), Sarcoma Collaborative Registry (SARCR), Melanoma Collaborative Registry (MELCR), Plasma Cell Dyscrasias Collaborative Registry (PDCR), Neuroendocrine Collaborative Registry (NETR), Non-Melanoma Skin Cancer Registry (NMSC) and Auxiliary Cancer Registry (ACR).

The iCaRe2 group elected to use a "confederation model", as opposed to a traditional registry or network model. The major advantages of a confederation model include the flexibility to use selected Centers for different research projects based on a Center's resources and expertise and the ability to have different strategies to address various research questions. A web-based registry iCaRe2 was developed and made available to any Center to participate in data collection and storage of cancer related data. The iCaRe2 provides a HIPAA compliant, secure, efficient and user-friendly mechanism for data and validation; utilization of standard vocabulary and data elements; and ad-hoc data reporting capabilities. The iCaRe2 serves as a collaboration platform for studies (including clinical trials) performed in centers with expertise in cancer biology, pathology, epidemiology, genetics, early detection, and patient care.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis/history of cancer
* Risk for developing cancer or suspicious clinical findings
* No history of cancer (normal control registry)
* Able to provide informed consent
* 19 years of age or older
* English or Spanish speaking individuals

Exclusion Criteria

* Unable to provide informed consent because of cognitive impairment
* Non-English or non-Spanish speaking individuals

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual who meets the eligibility criteria will be invited to participate in iCaRe2.
Sampling Method: Non-Probability Sample
Enrollment: 999999 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
Development and Implementation of a Web-based Cancer Collaborative Registry | 86 years
  This is a registry that will continue to accrue participants indefinitely.

SECONDARY OUTCOMES:
Procurement and Banking of Excess Biological Material for Future Analysis | 86 years
  This is a registry that will continue to accrue participants indefinitely.

OTHER OUTCOMES:
Collection and Banking of Blood, DNA, and Urine Samples for Future Studies | 86 years
  This is a registry that will continue to accrue participants indefinitely.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Fisher, MD, PhD, Principal Investigator — University of Nebraska
Locations (45):
- United States (45):
  - Advent Health, Greenwood Village, Colorado
  - Prospect Medical Hospital, Manchester, Connecticut
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Florida Hospital DeLand, DeLand, Florida
  - Florida Hospital FISH, Orange City, Florida
  - Florida Hospital Flagler, Palm Coast, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Covenant Medical Center, Inc, Waterloo, Iowa
  - Saint Luke's Cancer Instititute - South, Overland Park, Kansas
  - Northwest Hospital, Randallstown, Maryland
  - William E. Kahlert Regional Cancer Center, Westminster, Maryland
  - Holyoke Medical Center, Holyoke, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health-St. Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - St. Luke's Hospital of Duluth, Duluth, Minnesota
  - Lake Region Healthcare, Fergus Falls, Minnesota
  - Saint Luke's Cancer Institute, East, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City North, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Liberty, Liberty, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Heartland Regional Medical Center dba Mosaic Life Care, Saint Joseph, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Mary Lanning Healthcare, Morrison Cancer Center, Hastings, Nebraska
  - Faith Regional Health Services, Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Nebraska Methodist Health System, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - C.R. Wood Cancer Center, Glens Falls Hospital, Glens Falls, New York
  - Faxton St. Luke's Healthcare, Mohawk Valley, Utica, New York
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Essentia Health, Fargo, North Dakota
  - Trinity Hospital Cancer Care Center, Minot, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - Aultman Hospital, Canton, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rutland Regional Medical Center, Rutland, Vermont
  - Bellin Memorial Hospital, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All data and/or specimen request have to be made to the Principal Investigator of the center and follow the Human Subject Protection guidelines and policy.
Supporting Information: Study Protocol, ICF
Time Frame: as long as the registry is open
Access Criteria: Institutional Review Board approval to analyze data for separate study

REFERENCES:
- See also: icare2 website — http://icare2.unmc.edu